CLINICAL TRIAL: NCT06627543
Title: Effect of Enzyme Replacement Therapy on Cardiac Function in Children With Gaucher Disease Type 3
Status: Enrolling by invitation | Type: Observational
Sponsor: Noha Osman (Other)
Responsible Party: Sponsor-Investigator, Noha Osman, Lecturer, Assiut University
Organization: Assiut University (Other)
Other Study IDs: 04-2023-100034
Record Dates: First submitted 2024-09-29; First posted 2024-10-04 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2024-10

CONDITIONS: Gaucher Disease Type 3
MeSH Terms: conditions — Gaucher Disease | interventions — Caves

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Gaucher type patients
  Interventions: Diagnostic Test: echo

INTERVENTIONS:
Diagnostic Test: echo — echocardiographic

SUMMARY:
all cases confirmed diagnosis of Gaucher disease type 3 recieving enzyme replacement therapy at Assiut university hospital

DETAILED DESCRIPTION:
evaluate cardiac involvement in a group of GD type 3 patients, evaluate pulmonary hypertension and valvular involvement, compare the findings of basic echo before the start of replacement therapy as well as with healthy controls, to assess the effects of enzyme replacement therpay on the cardiac function.

ELIGIBILITY:
Inclusion Criteria:

* Any sex
* No age limit
* Gaucher disease type 3
* Receiving enzyme replacement therapy

Exclusion Criteria:

* Age18 years old
* Cases of gaucher type 1 and 2
* Other lipid storage disease

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: gaucher diseease type 3
Sampling Method: Non-Probability Sample
Enrollment: 44 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Evaluate Pulmonary Hypertension (PH) in Egyptian GD Type 3 Patients | 6 months
  To assess the presence and severity of pulmonary hypertension using echocardiography. Unit of Measure: mmHg (for systolic pulmonary artery pressure)
Evaluate Valvular Involvement in Egyptian GD Type 3 Patients | 6 months
  To assess the degree of valvular involvement, including stenosis or regurgitation, using echocardiography. Unit of Measure: Severity grading (mild, moderate, severe)

CONTACTS AND LOCATIONS:
Locations (1):
- Ahmed Mohammed Mohammed, Asyut, Egypt